CLINICAL TRIAL: NCT06063902
Title: Long-Term Opioid Therapy in Chronic Non-Cancer Pain: Risks and Benefits - A Prospective Cohort Study of Patients Treated in Specialized Pain Care
Brief Title: Long-Term Opioid Therapy in Chronic Non-Cancer Pain: Risks and Benefits
Status: Enrolling by invitation | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/376
Record Dates: First submitted 2023-01-12; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Chronic Non-Cancer Pain; Opioid Use Disorder
Keywords: Chronic pain; Chronic primary pain; Analgesics; Opioid; Opioid-use disorder; Work Ability; Health-related quality of life; Opioid-related risk behavior; Pain; Activity; Opioid-related complications
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study investigates long-term opioid treatment in patients with chronic non-cancer pain (CNCP). The study aims to prospectively identify predictive factors for work ability and for developing opioid use disorder (according to DSM-5) as well as predictive factors for pain, activity, and health-related quality of life.

It is hypothesized that certain biopsychosocial factors mapped in this study predict patterns of opioid use and the risk for developing OUD for patients with CNCP on long-term opioid therapy. Further, it is hypothesized that certain biopsychosocial factors mapped in this study predict the chance of improved work ability and other treatment benefits of long term opioid therapy in patients with CNCP.

DETAILED DESCRIPTION:
Chronic pain affects nearly 20% of the Swedish population. Pain from the musculoskeletal system together with psychiatric disorders are the chronic conditions that cost the most for the Swedish health care disability insurance and health care systems. Current knowledge suggests that chronic pain is maintained by changes in the nervous system together with psychological and social factors.

Opioids are known to be effective for acute and post-operative pain, and can be indispensable in palliative treatment of cancer pain. Long-term opioid therapy on the other hand is associated witg several risks, e.g., development of opioid dependence and opioid use disorder (OUD), and other opioid related complications including premature death. Clinical experience, qualitative and quantitative research suggest that some individuals with chronic pain do benefit from long-term opioid therapy in terms of clinical significant pain relief with only a low level of negative side-effects. However, evidence of change in functional outcomes and health related quality of life is ambiguous. Therefore, the role of long-term opioid therapy in chronic pain conditions remains debated and sometimes controversial.

In contrast to the well-established opioid epidemic in the U.S., little is known about the use of prescribed opioids in Sweden, and how this has developed during the last decade. The annual prevalence of opioid prescription did not change much during 2006-2017, but there were significant shifts in choice of opioids, with an increase in strong opioids e.g., oxycodone and morphine. Very little is known about what clinical consequences this shift might lead to.

The U-PAIN cohort study aims to examine patterns of prescribed opioid use, risks of adverse effects of long-term opioid therapy, and benefits of long-term opioid therapy, in a prospective clinical cohort.

The study aims to complete a broad bio-psycho-social characterization of the participants relevant to chronic pain. The study participants are followed over 5 years in order to study trajectories for patterns of opioid use, and predictive factors for opioid use disorder, work ability, pain severity and interference, and health-related quality of life.

At baseline, participants will be classified into 4 groups based on their current use of opioids:

1. No use
2. Short-term or intermittent use Criteria: short-term use defined as regular use of opioids for < 3 months or intermittent use as dosing up to 10 days/months (independent of time frame).
3. Long-term use with low to moderate doses Criteria: use of opioids for more > 3 months, more the 10 days/month and mean daily dose < 40 mg (oral morphine milligram equivalent dose (MEE) defined as low dose. Mean daily dose 40-100 mg MEE defined as high dose.
4. Long-term use with high doses Criteria: use of opioids for > 3 months. More than 100 mg MEE.

Main research questions for the cohort study are:

1. What characterizes patients without opioid use disorder at baseline compared to patients with mild, moderate or severe opioid use disorder respectively at baseline?
2. What variables predict their future:

   1. Patterns of opioid use and substance use disorder?
   2. Work ability, activity interference, quality of life and pain?

Potential predictors and co-variates include: (1) Individual factor and demographic variables (2) Pain characteristics, (3) Psychiatric co-morbidity and susceptibility for OUD, (3) Cognitive-behavioral variables, and (4) Physical functioning.

The objective is to identify the most salient predictors from each group and combine them into a final model with the best goodness of fit.

The four groups concerning patterns of opioid use will be statistically compared regarding key outcomes at baseline (opioid use disorders, work ability, activity interference, pain and HQoL)) by use of t-tests and chi-square tests. Logistic regression analyses will be applied for the study of predictors of opioid use, OUD, work ability, activity interference and pain. The dependent variables, e.g. OUD/no OUD will be regressed towards hypothetic predictors, grouped as described earlier, to end up with a final model including the most salient predictors from each group of variables. Multivariate regression models will be considered for continuous dependent variables.

In addition this clinical cohort will be open for other studies after ethical vetting, i.e. the cohort is unique and could contribute to further understanding of this population and hence should be open for further research.

ELIGIBILITY:
Inclusion Criteria:

1. Referral for a first visit to the Pain Centre of Uppsala University Hospital. The following
2. Competent in Swedish
3. Chronic Non-Cancer Pain (pain > 90 days)

Exclusion Criteria:

1. In active cancer treatment/Cancer-related pain
2. In palliative care
3. Need for interpreter
4. Cognitive impairment of magnitude that will prevent completion of study or ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe CNCP referred to secondary and tertiary pain care at the Uppsala University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Characterization and changes in opioid use disorder | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  As defined in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
  Measured by:
  Structured interview: Modified version of the Swedish Mini International Neuropsychiatric Interview, Part J (Substance use). Response format yes/no.
  Mild opioid use disorder = 2-3 symptoms Moderate opioid use disorder = 4-5 symptoms Severe opioid use disorder = 6 or more symptoms
Changes in work ability | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Self report. Work Ability Index (WAI). The questionnaire covers 7 dimensions:
  1. current work ability compared with lifetime best
  2. work ability in relation to the demands of the job
  3. number of diagnosed illnesses or limiting conditions
  4. estimated impairment owing to diseases/illnesses or limiting conditions
  5. amount of sick leave during the last year
  6. prognosis of work ability in 2 years' time
  7. psychological resources.
  The dimensions have different scores. A total index is computed ranging from 7 to 49, where higher scores indicate higher work ability. Individual items or sub-scales of WAI may also be used as outcome measures.

SECONDARY OUTCOMES:
Changes and patterns of opioid use (type of opioid, dose, and duration) | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  The Time Line Follow-Back (TLFB) Structured interview, calendar format, using 4 week intervals starting with the most recent complete week, week 1, working backward one week at a time recording days of use for each opioid.
Changes in pain severity and pain interference: The Brief Pain Inventory short-form (BPI-SF) | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Self report. The Brief Pain Inventory. Pain severity is measured with 4 items where worst, least, average, and current pain during the past week are scored. Each scale ranges from 0-10, where 0 = 'no pain' and 10 = 'pain as bad as can be'.
  Pain interference is measured with 7 items measuring how pain have interfered with the respondent's general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life during the last 24 ours. Each scale ranges from 0-10, where 0 = 'Does not interfere' and 10 = 'Interferes completely'.
  Higher scores indicate more pain severity and pain interference.
Changes in health related quality of life: EQ-5D-5L | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Self report. The EuroQoL - Five dimension (EQ-5D-5L). The five dimensions are: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of functioning: "1=no problems," "2=slight problems," "3=moderate problems," "4=severe problems," and "5=unable to"/ "extreme problems" for all dimensions that describe unique health states.The health states can be converted into index scores derived from population-based studies, that ranges from states worse than dead (<0) to 1 (full health), anchoring dead at 0.The EQ-5D questionnaire also includes a visual analog scale where perceived health status is rated with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Depressive symptoms | Baseline
  Self report: Patient Health Questionnaire - 9 (PHQ-9), Swedish version. 9 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. The first 9 items are summed to a sum score ranging from 0 to 27, where: 0-4 = no signs of depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression. Item 10 is reported as a single item where high scores indicate high interference with daily function.
Generalised Anxiety Disorder | Baseline
  Self report: Generalised Anxiety Disorder (GAD-7). 7 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. 1 item ranging from 0 ='not at all, to 3 = 'very disturbing'. The first 7 items are summed to a sum score ranging from 0 to 21, where: 0-4 = no signs of anxiety, 5-9 = mild GAD, 10-14 = moderate GAD, 15-21 = severe GAD. Item 8 is reported as a single item where higher score means higher interference.
Sleep | Baseline
  Self-report: The insomnia severity index (ISI) The ISI comprises 7 items that assess current (i.e., preceding 2 weeks) sleep problems. The first three items evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems. Subsequent items assess current sleep problem, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and amount of worry due to the current sleep problem. Items are rated on a five-point Likert scale ('0' representing none or not at all and '4' representing very much). Total scores range from 0 to 28, with higher combined scores indicating worse insomnia severity.
Pain self-efficacy | Baseline
  The Pain Self-Efficacy Questionnaire 2 (PSEQ-2), comprises 2 items that asses the participants beliefs about their ability to accomplish activities despite their pain: 'I can do some form of work, despite the pain. ("work" includes housework,paid and unpaid work)', and 'I can live a normal lifestyle, despite the pain'. Items are rated on a seven-point Likert scale ('0' not confident at all '6' Completelt confident). Total scores range from 0 to 12, with higher combined scores indicating stronger self-efficacy beliefs.
Experienced injustice | Baseline
  Self report: Injustice Experience Questionnaire (IEQ), Swedish version. IEQ measure the degree of experienced injustice following an injury. Respondents are asked to indicate on a five-point scale, ranging from 0 ='never, to 4 ='all the time'. The total score is calculated by adding the scores of each item. A total score is computed by summing the scores to all 12 items, ranging from 0-48 where higher scores indicate higher experience of injustice.
Fear of movement and reinjury | Baseline
  Self report, The Tampa Scale of Kinesiophobia-11 (TSK-11), Swedish version. 11 items ranging from 1 to 4 where 1 = 'does not agree at all', 4 = 'totally agree'. A total score is calculated ranging from 11 to 44 where higher scores indicate higher fear of movement/kinesiophobia.
Catastrophizing - The Pain Catastrophizing Scale (PCS) - Swedish version. | Baseline
  Self report, self-administered form. The Pain Catastrophizing Scale (PCS) - Swedish version. 13 items, ranging from 0 to 4 where 0 = 'not at all', 4 = 'all the time'. A total score is calculated ranging from 0 to 52 where higher scores indicate higher catastrophizing.
Changes in life habits | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
  Self-report. The Lifestyle questionnaire by the Swedish National Board of Health. Assesses physical activity and sedentary (duration in minutes and intensity), tobacco use (any use, tobacco cessation= stopped using> 6 month ago or stopped< than 6 months, and amount), diet (eating vegetables, fruit/berries, fish or shellfish, and candy/cookies; twice/day, once/day, couple of times/week, once/week, couple of times/month or less. Breakfast; every day, almost every day, few days/week, one/week or less) and alcohol use (any use, occasions/week and amount).
Alcohol Use | Baseline
  Self report: Alcohol Use Disorder Identification Test (AUDIT) Swedish version, a 10-item measure of past-year harmful and hazardous alcohol use. The AUDIT addresses three conceptual domains: alcohol consumption (three items), alcohol-related problems (four items), and adverse psychological reactions (three items). The first 8 items are scored on a 5-point scale ranging from 0 to 4, and the last two are scored on a 3-point scale with values 0, 2, and 4. The total score ranges from 0-40 with cut-off values of 8 and 6 points for men and women respectively indicate hazardous alcohol use and a score of ≥19, indicates alcohol-related problems including dependence.
Illicit drug use | Baseline
  Self report. The Drug Use Disorder Identification test (DUDIT) Swedish version,an 11-item screening instrument developed to identify non-alcohol drug use patterns and drug-related problems. The first nine items are scored on a 5-point scale ranging from 0 to 4, and the last two are scored on a 3-point scale with values 0, 2, and 4. Thus, scores range from 0-44 with higher scores indicating a more severe drug problem, with cut-off values of 4 and 2 points for men and women respectively indicate hazardous drug use.
Pain classification | Baseline
  International classification of disease (ICD-11).
Personality traits | Baseline
  Self report. Swedish universities scale of personality (SSP), an instrument developed to measure personality traits intended to be markers for various neurobiological processes related to vulnerability to mental illness. It consists of 91 items that generates 13 different scales. For all items the respondent fill in one of four possible answer alter; not true at all, does not match particularly well, agree somewhat, exactly right. Each of the 13 scales represent relevant personality aspects and are as follow; Somatic trait anxiety (STA), Psychic trait anxiety (PsTA), Stress susceptibility (SS), Lack of assertiveness (LA), Detachment (D), Embitterment (E), Mistrust (M), Physical trait aggression (PhTA), Verbal trait aggression (VTA), Adventure seeking (AS), Impulsiveness (I), Social desirability (SD), and Trait irritability (TI). SSP has also been factor-analysed into three major dimensions, Neuroticism, Aggressiveness and Extraversion.
Attention-deficit hyperactivity disorder (ADHD) symptoms | Baseline
  Self report. ADHD Self-Report Scale (ASRS v.1.1) includes 18 items of recent DSM-IV Criterion A symptoms of adult ADHD. Respondents are asked how often a symptom has occurred over the past 6 months on a scale ranging from 0 to 4 (never, rarely, sometimes, often and very often).
Life-time experience of traumatic events | Baseline
  Self-report. the Life Events Checklist (LEC) consists of 16 items inquiring about the experience of 16 different potentially traumatic events (PTE) known to result in PTSD or other posttraumatic difficulties. For each PTE, respondents rate their experience of that event on a 5-point nominal scale (1 = happened to me, 2 = witnessed it, 3 = learned about it, 4 = not sure, and 5 = does not apply).
Walk speed | Baseline
  Physical functional test. 10 meters test of walking
Balance | Baseline
  Physical functional test.The Mini Balance Evaluation Systems Test (mini-BESTest) consist of 14 item measuring dynamic balance. Each item is scored on a 3-category ordinal scale from 0 (unable or requiring help to perform) to 2 (normal) with a total score from 0 to 28.
Substance use and substance use disorder | Baseline
  Structured interview: Modified version of the Swedish Mini International Neuropsychiatric Interview, Part J (Substance use). The M.I.N.I (J) assesses eight categories of substances, including both prescribed medications and illicit substances: opioids (heroin and opium as a separate category), stimulants, cocaine, hallucinogens, inhalants, marijuana, and benzodiazepines. The substance use disorder section was modified to assess current as well as life-time drug use, and medical as well as non-medical use. Response format yes/no.
  Substance use disorder defined in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
  Mild substance use disorder = 2-3 symptoms Moderate substance use disorder= 4-5 symptoms Severe substance use disorder = 6 or more symptoms
Explorative identification of change in biomarkers | Baseline
  Biomarkers will be explored by use of the OLINK (name of brand) panel which enables analysis of 92 inflammation-related protein biomarkers.
Experienced effect of treatment/Global goal achievement | 1 year
  Self report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.
Experienced effect of treatment/Global goal achievement | 2 year
  Self report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.
Experienced effect of treatment/Global goal achievement | 3 year
  Self report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.
Experienced effect of treatment/Global goal achievement | 4 year
  Self report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.
Experienced effect of treatment/Global goal achievement | 5 year
  Self report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.

OTHER OUTCOMES:
Sick-leave | Baseline
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Sick-leave | 1 year
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Sick-leave | 2 year
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Sick-leave | 3 year
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Sick-leave | 4 year
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Sick-leave | 5 year
  Register data. Average sick leave according to the Swedish Social Insurance register, defined as net days.
Prescribed drugs | Baseline
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.
Prescribed drugs | 1 year
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.
Prescribed drugs | 2 year
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.
Prescribed drugs | 3 year
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.
Prescribed drugs | 4 year
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.
Prescribed drugs | 5 year
  Register data. Drug outtake according to the drug register held by the Swedish National Board of Health.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Professor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala Univeristy Hospital, Uppsala, Sweden